CLINICAL TRIAL: NCT02809482
Title: Pilot Study to Examine the Impact of Overfeeding on Peripheral Clock Gene Expression in Humans
Brief Title: White Adipose Tissue Clocks and High Calorie Feeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 15-1570; UL1TR001082 (NIH)
Record Dates: First submitted 2015-12-07; First posted 2016-06-22 (Estimated); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Healthy
Keywords: Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eucaloric Feeding (Other)
  Interventions: Other: Eucaloric feeding
- Overfeeding (Other)
  Interventions: Other: Overfeeding

INTERVENTIONS:
Other: Eucaloric feeding — 3 days of a diet designed to maintain energy balance
  Arms: Eucaloric Feeding
Other: Overfeeding — 3 days of a diet designed to induce a 40% positive energy balance
  Arms: Overfeeding

SUMMARY:
Peripheral tissues (e.g. liver, adipose, muscle) express self-sustained circadian clocks that coordinate daily metabolic rhythms. The timing of clock rhythms in peripheral tissues is highly sensitive to feeding-fasting signals across the sleep-wake transition. Nutritional insults such as high fat overfeeding (HF-OF) have been shown to attenuate clock gene expression in peripheral tissues resulting in a deleterious re-programming of the circadian metabolome. Studies in humans have only superficially investigated how the circadian clock machinery is impacted by nutritional signals. The overall goal of this pilot project is to take the first steps toward developing translational methods to investigate links between changes in energy flux and the circadian system in human tissues. Using an innovative ex vivo cell culture approach the investigators will examine the impact of 3-days of HF-OF compared to eucaloric (EU) feeding on the expression of core clock genes in human subcutaneous adipose tissue (SAT). The Investigators hypothesize that compared to EU, the amplitude of clock gene expression in SAT measured over 24hrs will be attenuated following short-term HF-OF. This pilot project will serve as a launch point for designing future studies into the effects of diet and exercise on the circadian control of metabolism in adipose tissue depots as well as other tissues (e.g. muscle).

ELIGIBILITY:
Inclusion Criteria:

* males and females aged 20-35 yr;
* BMI 25-35 kg/m2 and weight stable (±2kg in past 2mo);
* non-smoker;
* sedentary to moderately active (≤3 days of exercise per week ≤30 min of exercise per session);
* sleeping pattern of >7 hours to 9.25 hrs of sleep/night.
* subjects will be asked to identify themselves as regular consumers of 3 balanced meals per day by answering the question: "Do you eat breakfast, lunch, and dinner on ≥ 5 days per week?"

Exclusion Criteria:

* Smoker (current or within the previous 3 months);
* Use any medication that could affect lipid metabolism, insulin signaling, or sleep;
* Pregnant women will not be enrolled in the study;
* Have a job that involves shift work;
* Dwelling below Denver altitude (1,600 m) a year prior to testing;
* Travel across more than one time zone 3 wk before a study;
* chronic health conditions such as diabetes, hyper or hypothyroidism, renal or liver disease, anemia, or cancer;
* Regularly go to sleep after midnight;

  o Subjects will be excluded if they are identified as having night eating syndrome (at least 25% of food intake is consumed after the evening meal and/or at least two episodes of nocturnal eating per week);
* Allergy to lidocaine or similar compound;
* Have one or more of the following out-of-range values measured on a fasting blood sample:

  * glucose > 110 mg/dl,
  * thyroid stimulating hormone <0.5 or >5.0 µU/ml.
* Subjects who may be:

  * anemic (hemoglobin < 14.5 g/dl men, <12.3 g/dl women ),
  * have abnormal liver function tests (alanine amino transferase > 47 U/l, aspartate aminotransferase, > 47 U/l, alkaline phosphatase <39 or >117 U/l) or creatinine (>1.1 mg/dl).

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Expression of clock genes in adipose tissue. | Measured through study completion, an average of 4 weeks.
  Gene expression measured at two time points from abdominal fat.

SECONDARY OUTCOMES:
Gene expression of key cellular fuel sensors thought to be controlled. and/or influenced by peripheral clocks | Measured through study completion, an average of 4 weeks.
  Gene expression measured at two time points from abdominal fat.
Expression of clock genes in blood monocytes. | Measured through study completion, an average of 4 weeks.
  Gene expression measured at two time points from abdominal fat.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bessesen, MD, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoo SH, Yamazaki S, Lowrey PL, Shimomura K, Ko CH, Buhr ED, Siepka SM, Hong HK, Oh WJ, Yoo OJ, Menaker M, Takahashi JS. PERIOD2::LUCIFERASE real-time reporting of circadian dynamics reveals persistent circadian oscillations in mouse peripheral tissues. Proc Natl Acad Sci U S A. 2004 Apr 13;101(15):5339-46. doi: 10.1073/pnas.0308709101. Epub 2004 Feb 12. PMID 14963227
- [Background] Oosterman JE, Kalsbeek A, la Fleur SE, Belsham DD. Impact of nutrients on circadian rhythmicity. Am J Physiol Regul Integr Comp Physiol. 2015 Mar 1;308(5):R337-50. doi: 10.1152/ajpregu.00322.2014. Epub 2014 Dec 17. PMID 25519730
- [Background] Eckel-Mahan KL, Patel VR, de Mateo S, Orozco-Solis R, Ceglia NJ, Sahar S, Dilag-Penilla SA, Dyar KA, Baldi P, Sassone-Corsi P. Reprogramming of the circadian clock by nutritional challenge. Cell. 2013 Dec 19;155(7):1464-78. doi: 10.1016/j.cell.2013.11.034. PMID 24360271
- [Background] Pivovarova O, Jurchott K, Rudovich N, Hornemann S, Ye L, Mockel S, Murahovschi V, Kessler K, Seltmann AC, Maser-Gluth C, Mazuch J, Kruse M, Busjahn A, Kramer A, Pfeiffer AF. Changes of Dietary Fat and Carbohydrate Content Alter Central and Peripheral Clock in Humans. J Clin Endocrinol Metab. 2015 Jun;100(6):2291-302. doi: 10.1210/jc.2014-3868. Epub 2015 Mar 30. PMID 25822100
- [Derived] Rynders CA, Morton SJ, Bessesen DH, Wright KP Jr, Broussard JL. Circadian Rhythm of Substrate Oxidation and Hormonal Regulators of Energy Balance. Obesity (Silver Spring). 2020 Jul;28 Suppl 1(Suppl 1):S104-S113. doi: 10.1002/oby.22816. Epub 2020 May 28. PMID 32463976